CLINICAL TRIAL: NCT00537160
Title: The Impact of a Diet and Exercise Program in Overweight Pediatric Patients During Burn Rehabilitation
Brief Title: Diet and Exercise in Overweight Children Postburn
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Michele Gottschlich, Research Dietitian, Shriners Hospitals for Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-04-26-01
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Obesity; Burns
Keywords: Pediatrics
MeSH Terms: conditions — Obesity; Burns | interventions — Behavior Therapy; Nutrition Assessment; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Behavior modification, Nutrition Education, Exercise

SUMMARY:
Examine clinical results of an interdisciplinary weight management program that includes medical evaluation, nutrition counseling, exercise, and behavioral interventions.

ELIGIBILITY:
Inclusion Criteria:

* 10-18 years old
* BMI > or = 95th percentile
* > 1 year postburn and out of pressure garments
* Live within 100 minle radius of SHC
* Informed consent and HIPPA form signed
* Parent/guardia willing to make time commitment

Exclusion Criteria:

* Undergone major surgery in the 4 months prior to start of program or have any major surgery planned in 2 year time frame
* Physical/health condition that precludes regular exercise
* Significant mental health diagnosis
* Advised by MD not to exercise
* Thyroid disease, routine steroid use,pregnancy
* Unable to understand the instructions/content of program

Ages: 10 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2006-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
BMI | 12 and 24 months following intervention

SECONDARY OUTCOMES:
fitness level | 12 and 24 months following intervention

CONTACTS AND LOCATIONS:
Overall Officials: Michele M Gottschlich, PhD, RD, CNSD, Principal Investigator — Shriners Hospital for Children